CLINICAL TRIAL: NCT00140933
Title: A Randomized, Double-Blind, 7-Day Study of the Efficacy and Safety of Rofecoxib Versus Placebo and Diclofenac in Patients With Acute Painful Rotator Cuff Syndrome
Brief Title: A Study to Evaluate Rofecoxib Versus Placebo and Diclofenac in Patients With Acute Painful Rotator Cuff Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005_056
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2006-12-05 (Estimated); Status verified 2006-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — rofecoxib

INTERVENTIONS:
Drug: MK0966; rofecoxib
Drug: Comparator: diclofenac, placebo

SUMMARY:
Comparing the short-term efficacy of rofecoxib versus placebo. Patients receive rofecoxib or placebo or diclofenac and fill out a patient diary on daytime pain severity during daily activities, night pain severity, and acetaminophen/paracetamol intake.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 59 with acute painful rotator cuff syndrome.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 274
Dates: Start 2003-04

PRIMARY OUTCOMES:
Pain during daily activities assessed by a Numerical Rating Score (NRS)

SECONDARY OUTCOMES:
Functional impairment evaluated using Neer's functional index.
Global assessment of disease activity by the patient with a NRS.
Intensity of night pain evaluated by NRS.
Rescue treatment take during the study duration.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Laboratoires Merck Sharp & Dohme - Chibret, Paris, France

REFERENCES:
- [Derived] Jones P, Lamdin R, Dalziel SR. Oral non-steroidal anti-inflammatory drugs versus other oral analgesic agents for acute soft tissue injury. Cochrane Database Syst Rev. 2020 Aug 12;8(8):CD007789. doi: 10.1002/14651858.CD007789.pub3. PMID 32797734